CLINICAL TRIAL: NCT06984055
Title: Diagnostic Accuracy of Deep Learning-Assisted Multimodal Endocytoscopy for Superficial Esophageal Neoplasia and Precancerous Lesions: A Multicenter ，Prospective Study
Brief Title: Diagnostic Accuracy of Endocytoscopy for Superficial Esophageal Neoplasia
Status: Enrolling by invitation | Type: Observational
Sponsor: Changhai Hospital (Other)
Collaborators: Ruijin Hospital (Other); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); the Tenth People's Hospital affiliated to Tongji University (Unknown); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); First Affiliated Hospital of Zhejiang University (Other); Sir Run Run Shaw Hospital (Other); The Second Hospital of Nanjing Medical University (Other); Jiangsu Province Hospital of Traditional Chinese Medicine (Other); The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Luowei Wang, MD, Clinical Professor, Changhai Hospital
Other Study IDs: DAESEN
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Esophageal Cancer, Squamous Cell
Keywords: Endocytoscopy; Esophageal Neoplasia; Precancerous Lesions; Deep Learning
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In recent years, endocytoscopy (EC) has undergone rapid development as an advanced endoscopic technique. Characterized by real-time histological imaging and detection capabilities, EC enables visualization of living cells in the digestive mucosal layer through methylene blue staining via the endoscopic instrument channel. This technology provides ultra-magnified endocytoscopic images, allowing for identification of key cellular features including epithelial cell morphology and the shape of methylene blue-stained epithelial nuclei, thereby facilitating clear in vivo observation of microstructural characteristics in mucosal tissues - a technique commonly referred to as "optical biopsy". However, current clinical application of EC in China remains limited due to insufficient practical experience and the absence of standardized diagnostic criteria for image interpretation. This study aims to comprehensively evaluate the diagnostic accuracy of domestically developed high-magnification electronic upper gastrointestinal endoscopy for esophageal carcinoma and precancerous lesions, using histopathology as the gold standard. The research objectives include establishing standardized diagnostic evaluation protocols and clarifying the clinical value of this technology through systematic validation.

ELIGIBILITY:
Inclusion Criteria:

1.Patients diagnosed with superficial esophageal squamous cell carcinoma or high-grade intraepithelial neoplasia (HGIN) through endoscopic and pathological biopsy examinations, scheduled for endoscopic submucosal dissection (ESD); 2.Patients with esophageal squamous low-grade intraepithelial neoplasia (LGIN) confirmed by endoscopic and biopsy histopathological examinations within the preceding six months; 3. Patients exhibiting esophageal focal lesions detected during painless upper gastrointestinal endoscopy requiring pathological biopsy.

Exclusion Criteria:

1. Patients aged <18 years or >80 years;
2. Lesions located at the gastroesophageal junction with clinical suspicion of adenocarcinoma or precancerous lesions;
3. Patients with contraindications to sedated/anesthetized upper gastrointestinal endoscopy;
4. Patients with coagulation disorders;
5. Patients with a history of hypersensitivity to relevant medications (including anesthetics or methylene blue);
6. Patients presenting dysphagia or gastrointestinal obstructive symptoms, or those with suspected/confirmed digestive tract obstruction, stenosis, or fistulae;
7. Patients declining to provide informed consent for study participation, or any other circumstances deemed by investigators to preclude eligibility.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population who underwent endocytoscopy due to related symptoms from April 2025 to December 2026
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | 10 minutes
  sensitivity and specificity

CONTACTS AND LOCATIONS:
Overall Officials: Wang Luowei, Principal Investigator — Changhai hosipital, Shanghai
Locations (1):
- Changhai hosipital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No